CLINICAL TRIAL: NCT01401179
Title: Randomized Phase III Trial of Cefazolin or Combination of Cefazolin and Erythromycin or Cefazolin and Clarithromycin in Women With Preterm Premature Rupture of the Membranes
Brief Title: Antibiotics Study in Preterm Premature Rupture of the Membranes
Acronym: PPROM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Soo-young Oh, M.D. PhD, Department of Obstetrics and Gynecology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-04-003
Record Dates: First submitted 2011-07-19; First posted 2011-07-25 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-07

CONDITIONS: Preterm Premature Rupture of the Membranes
Keywords: Preterm Premature Rupture of Fetal Membranes; antibiotic therapy
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Fetal Membranes, Premature Rupture | interventions — Cefazolin; Erythromycin; Clarithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- cefazolin (Active Comparator)
  Interventions: Drug: cefazolin, erythromycin, clarithromycin
- cefazolin plus erythromycin (Active Comparator): cefazolin, erythromycin
  Interventions: Drug: cefazolin, erythromycin, clarithromycin
- cefazolin plus clarithromycin (Active Comparator)
  Interventions: Drug: cefazolin, erythromycin, clarithromycin

INTERVENTIONS:
Drug: cefazolin, erythromycin, clarithromycin — Antibiotics regimen was one of cefazolin or cefazolin plus erythromycin or cefazolin plus clarithromycin. Intravenous 1g cefazolin was given every 6 hours after negative result skin test for allergic reaction. With cefazolin plus erythromycin group or cefazolin plus clarithromycin, cefazolin was given with same protocol and 250mg oral erythromycin every 6 hours or 500mg oral clarithromycin every 12 hours was added. All antibiotics were given for 7 days or until delivery.

SUMMARY:
The purpose of this study is to compare the efficacy on maternal infection, chorioamnionitis and neonatal morbidity and mortality, and to review the evidence and provide recommendations on the use of antibiotics in PPROM.

DETAILED DESCRIPTION:
Despite major advances in perinatal care, preterm delivery is still the predominant cause of perinatal mortality and a major cause of neurological morbidity and mortality. Although the determinants of preterm labor and delivery are uncertain, evidence suggests intrauterine infection is a contributing factor. Antibiotic therapy for women in preterm premature rupture of membranes has been a routine practice. However the optimal regimen remains unclear and the choice of latency antibiotic regimen is at the discretion of admitting physician. The group 1 is treated only with cefazolin (1.0mg iv every 6 hours for 7 days). The group 2 is given a combination of cefazolin(1.0mg iv every 6 hours for 7 days) and erythromycin(250mg p.o. four times a day for 7 days). In group 3, clarithromycin (500mg p.o. 4 times a day for 7 days) was treated with cefazolin(1.0mg iv every 6 hours for 7 days). This study is designed to compare the efficacy on maternal infection, chorioamnionitis and neonatal morbidity and mortality and to review the evidence and provide recommendations on the use of antibiotics, especially by comparing the combination regimen in PPROM.

ELIGIBILITY:
Inclusion Criteria:

* PPROM, PA 23+0~33+0wks
* ROM <48 hrs before randomization
* singleton
* Cervical dilatation <3cm
* uterine contraction less than 4 times per 1 hr

Exclusion Criteria:

* Major fetal malformation
* Multifetal pregnancy
* Rupture of the membrane >8hrs before randomization
* Prior antibiotics use at local clinic before referral
* Vaginal bleeding
* IIOC (incompetent internal os of cervix)
* Placenta previa
* Gestational diabetes or overt diabetes
* Hypertensive disorders in pregnancy
* Liver cirrhosis
* Acute renal failure
* IUGR(Intrauterine growth restriction)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Neonatal composite morbidity | Participants will be followed for duration of hospital day after delivery, an expected average of 8 weeks.
  1. respiratory distress syndrome(RDS)
  2. bronchopulmonary dysplasia(BPD)
  3. intraventricular hemorrhage(IVH,≥grade 3)
  4. retinopathy of prematurity(ROP,≥grade 3)
  5. necrotizing enterocolitis(NEC,≥stage 2)
  6. proven neonatal sepsis

SECONDARY OUTCOMES:
the incidence of abnormal brain sonography | Participants will be followed for duration of hospital day after delivery, an expected average of 8 weeks.
infantile neurologic outcome | at 6 months and 1 year of corrected age
  The outcome was evaluated in five sub-domains (development, neurologic examination, Bayley Scales of Infant Development-II, vision, and hearing). The final outcome scale was divided into normal, mild, moderate, and severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Young Oh, M.D., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical center, Seoul, South Korea